CLINICAL TRIAL: NCT04624698
Title: iStent Inject Trabecular Micro-Bypass System New Enrollment Post-Approval Study
Brief Title: iStent Inject New Enrollment Post-Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG2M-105-PASN
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma, Open-Angle; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Implantation (Experimental): Subjects will undergo cataract surgery and then implantation of the iStent Inject trabecular micro-bypass device.
  Interventions: Device: iStent Inject Implantation

INTERVENTIONS:
Device: iStent Inject Implantation — Subjects will be implanted with the iStent Injection Micro-Bypass device

SUMMARY:
Study to evaluate the rate of clinically relevant complications associated with iStent inject placement in the post-market setting.

DETAILED DESCRIPTION:
To evaluate the rate of clinically relevant complications associated with iStent inject placement and stability, as determined at 36 months in the postmarket setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 22 years of age
2. Mild to moderate primary open-angle glaucoma
3. Scheduled to undergo cataract surgery
4. Able and willing to attend scheduled follow-up exams for three years postoperatively
5. Able and willing to provide written informed consent on the IRB approved Informed Consent Form

   Operative Inclusion Criterion:
6. Successful, uncomplicated cataract surgery

Exclusion Criteria:

1. Angle closure glaucoma
2. Traumatic, malignant, uveitic, or neovascular glaucoma or discernible congenital anomalies of the anterior chamber angle
3. Retrobulbar tumor, thyroid eye disease, Sturge-Weber Syndrome or any other type of condition that may cause elevated episcleral venous pressure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
iStent inject placement and stability | 36 Months
  The rate of clinically relevant complications associated with iStent inject placement and stability

SECONDARY OUTCOMES:
Sight-threatening adverse events | 36 Months
  Rate of occurrence of sight-threatening adverse events

OTHER OUTCOMES:
Other adverse events | 36 Months
  Rate of other adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Eye Doctors of Arizona, PLLC, Phoenix, Arizona
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Glaucoma Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No